CLINICAL TRIAL: NCT00519415
Title: This Study is to Apply the Tongue Force to Correct the Dentofacial Deformities
Brief Title: Comparative Results of Maxillary Deficiency Treatment by Tongue Plate and Facemask in Growing Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Mahkameh Mirkarimi, Shaheed Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13425678; 1234567
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Maxillary Deficiency
Keywords: Tongue plate; Facemask; class III maxillary deficiency; orthodontic angle class three
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Other: Tongue plate
- B (Experimental)
  Interventions: Other: Facemask

INTERVENTIONS:
Other: Tongue plate — A functional appliance use for maxillary protraction.It has two adams clasp and two C clasp to retained the appliance and long palatal plate in the canine area which cages the tongue and transfer the force of the tongue during physiological activity to the upper arch. It has posterior bite plate and middle screw for maxillary expansion.It should be used all the time except meal time and brushing the teeth,the acrylic appliance makes specifically for the patient.
  Other Names: tongue appliance
  Arms: A
Other: Facemask — An extraoral appliance use for treatment of maxillary deficiency in growing patients.It takes anchorage from chin and forehead, it has removable intraoral appliance with hooks for elastics that exerted a force of 300 gr.It should be used 14 hours a day.
  Other Names: Reverse pull headgear
  Arms: B

SUMMARY:
A new appliance will be used to transfer the tongue force during its physiological activity to advance the nasomaxillary complex; this method will be compared with the traditional method which uses a Facemask appliance.

DETAILED DESCRIPTION:
The above method will be compared with traditional one which uses the Facemask in combination with an intra-oral appliance.

ELIGIBILITY:
Inclusion Criteria:

* Growing patients
* Class III with maxillary deficiency

Exclusion Criteria:

* Previous orthodontic treatment
* Un cooperative patients

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Cephalometric angles and clinical features | At least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lida Toomarian, Study Chair — Shaheed Beheshti dental school; Rahman Showkatbakhsh, Study Director — Shaheed Beheshti dental shool; Mahkameh Mirkarimi, Principal Investigator — Shaheed Beheshti dental shool
Locations (1):
- Shaheed Beheshti dental school, Tehran, Iran